CLINICAL TRIAL: NCT04608604
Title: Mobility in Atypical Parkinsonism: a Randomized Trial of Physiotherapy
Brief Title: Mobility in Atypical Parkinsonism: a Trial of Physiotherapy
Acronym: Mobility_APP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Victoria Sidoroff (Other)
Collaborators: University of Lausanne Hospitals (Other); Medical University Innsbruck (Other); University of Luxembourg (Other); Friedrich-Alexander-Universität Erlangen-Nürnberg (Other); Regional Hospital of Bolzano (Other); Ecole Polytechnique Fédérale de Lausanne (Other); University Hospital Erlangen (Other); Reha Rheinfelden (Other); Klinik Lengg, Zurich (Other)
Responsible Party: Sponsor-Investigator, Victoria Sidoroff, Study Investigator, Department of Neurology, Medical University of Innsbruck, Universitätsklinik für Neurologie, Innsbruck
Organization: Universitätsklinik für Neurologie, Innsbruck (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1290/2020
Record Dates: First submitted 2020-10-19; First posted 2020-10-29 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Multiple System Atrophy, Parkinson Variant (Disorder); Parkinson Disease; Progressive Supranuclear Palsy
MeSH Terms: conditions — Multiple System Atrophy; Parkinson Disease; Supranuclear Palsy, Progressive | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physiotherapy 1 (Active Comparator)
  Interventions: Other: Physiotherapy
- Physiotherapy 2 (Active Comparator)
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Patients will be randomized in either physiotherapy 1 or physiotherapy 2. Physiotherapy programs are individually tailored based on a structured standardized series. In order to not unblind potential participants, detailed description of both interventions will be provided after recruitment has been finished.

SUMMARY:
Patients with atypical parkinsonism often show gait and mobility impairment manifesting in early disease stages.

In order to maintain mobility and physical autonomy as long as possible for these patients, we will examine the effect of two types of physiotherapy in patients with multiple system atrophy (MSA), progressive supranuclear gaze palsy (PSP) and idiopathic Parkinson's disease (IPD).

The study is divided into an ambulant daily in-patient physiotherapy phase, followed by a home-based training phase. At the beginning and the end of the study, the patients daily activity will be recorded for one week using Physical Activity Monitoring (PAM) sensors.

The aim of this double-blind, randomized-controlled study is to determine effective physiotherapy in patients with atypical parkinsonian syndromes in order to maintain mobility for as long as possible.

DETAILED DESCRIPTION:
Patients with Parkinson's disease often show gait impairment and reduced mobility over the disease course. Rare atypical forms of parkinsonism, like multiple system atrophy (MSA) or progressive supranuclear gaze palsy (PSP) develop these features in early disease stages. The reduced mobility and increased time spent in sitting or lying posture leads to loss of physical independence and increased mortality. Since MSA and PSP can currently only be treated symptomatically, a long lasting independence and mobility is therefore of great importance.

A positive effect has already been shown in a few studies on specific physiotherapy in patients with idiopathic Parkinson's disease (IPD), and some small studies also give us an evidence that physiotherapy in atypical parkinsonism can improve mobility.

The Mobility_APP study examines the effect of two types of physiotherapy in patients with MSA, PSP and IPD. The participants are initially assigned to a type of therapy and they learn specific exercises with a physiotherapist every day for two weeks. These exercises will then be continued independently at home for another five weeks. Regular checks in the study center ensure a precise examination of the physical condition, quality of life and gait pattern. The latter will be objectively analyzed with the help of sensors that are worn on the participant's shoes. In addition, before the start and at the end of the study, the participants are also monitored for one week at home using shoe sensors in order to reflect the natural conditions of the patients.

During the entire study, neither the participant nor the study investigator knows what type of therapy is being used in order to guarantee an unbiased analysis (double blinding).

The aim of this double-blind, randomized-controlled study is to determine effective physiotherapy in patients with atypical parkinsonian syndromes in order to maintain mobility for as long as possible. If the exercises learned during physiotherapy can be continued regularly at home and can improve mobility, this means a big step towards autonomous therapy. Frequent visits to therapists can be reduced and sufficient and effective independent therapy can still be carried out during times of crisis or phases with increased motor impairment.

The project is kindly supported by the Fund for the Promotion of Scientific Research (FWF). Together with the German Research Foundation (DFG) and Swiss National Science Foundation (SNF) in Switzerland this project can be carried out internationally in cooperation with renowned centers for neurological and sensor-based research.

ELIGIBILITY:
Inclusion Criteria:

* The subject is willing and able to give written informed consent
* The patient is able to tolerate all study visits including daily physiotherapy and home training.
* Patients similar with regard to age and sex with probable/possible MSA-P according to rev. Gilman criteria OR probable/possible PSP-RS according to MDS-PSP criteria OR PD according to MDS-PD criteria.
* Stable antiparkinsonian and Anti-OH medication 4 weeks prior to study entry.

Exclusion Criteria:

* Co-morbidities that influence the clinical presentation of parkinsonian symptoms (as judged by the enrolling investigator).
* Participation in other clinical trials that might influence the impact of the trial intervention (as judged by the enrolling investigator)
* H&Y Staging score greater than or equal to 4
* Change of antiparkinsonian and anti-OH medication 4 weeks prior to the interventional trial.
* Secondary cause of autonomic failure or parkinsonism (e.g. diabetic autonomic neuropathy, bladder surgery, drug-induced or vascular parkinsonism, etc.)
* Dementia according to DSM-V.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Sensor-based analysis | Baseline to week 7
  Gait speed

SECONDARY OUTCOMES:
Clinical Rating scale | Baseline to week 7
  Movement Disorder Society - Unified Parkinson's Disease Rating Scale - MDS-UPDRS III (0-132 points, higher scores indicate higher motor impairment)
Sensor-based analysis | Baseline to week 7
  Stride length
PAM Secondary outcome | Baseline to week 7
  Number of steps per day

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sidoroff V, Moradi H, Prigent G, Jagusch F, Teckenburg I, Asalian M, Hergenroeder-Lenzner N, Giraitis M, Schoenfeldt-Reichmann ET, Ndayisaba JP, Goebel G, Seppi K, Ionescu A, Krismer F, Benninger D, Winkler J, Eskofier BM, Klucken J, Aminian K, Wenning G, Sapienza S, Gassner H, Raccagni C; MobilityAPP Study Group. Moving beyond the hospital: in-depth characterization of daily-life mobility in patients with atypical Parkinsonian disorders. NPJ Parkinsons Dis. 2026 Jan 12. doi: 10.1038/s41531-025-01242-2. Online ahead of print. PMID 41526364
- [Derived] Raccagni C, Sidoroff V, Paraschiv-Ionescu A, Roth N, Schonherr G, Eskofier B, Gassner H, Kluge F, Teatini F, Seppi K, Goebel G, Benninger DH, Aminian K, Klucken J, Wenning G. Effects of physiotherapy and home-based training in parkinsonian syndromes: protocol for a randomised controlled trial (MobilityAPP). BMJ Open. 2024 May 1;14(5):e081317. doi: 10.1136/bmjopen-2023-081317. PMID 38692728